CLINICAL TRIAL: NCT03461263
Title: Trans-perineal Pumpkin Seeds Phonophoresis as an Adjunct Treatment for Chronic Non-bacterial Prostatitis
Brief Title: Effect of Pumpkin Seeds Phonophoresis on Chronic Non-bacterial Prostatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahlia University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Dr Sayed Tantawy, Associate Professor, Ahlia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: No: P. T. REC/ 012/001810
Record Dates: First submitted 2018-03-04; First posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Chronic Non-bacterial Prostatitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Group A, wherein patients received phonophoresis treatment using pumpkin seeds oil; Group B, where members of the group received trans-perineal continuous low-intensity ultrasound; and Group C, in which the participant received placebo low- intensity ultrasound. All of The three groups of the organized trail received their corresponding treatment daily up-to 3 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): phonophoresis treatment using pumpkin seeds oil
  Interventions: Other: phonophoresis treatment using pumpkin seeds oil
- Group B (No Intervention): Low intensity Ultrasound
- Group C (No Intervention): Placebo Low intensity Ultrasound

INTERVENTIONS:
Other: phonophoresis treatment using pumpkin seeds oil — phonophoresis treatment using pumpkin seeds oil
  Arms: Group A

SUMMARY:
It has been observed that out of all visits to the clinics by the young and middle age men for grievances including the genital and urinary frameworks, about 25% of the visits account for Prostatitis. A significant number of men, aged less than 50, visits to urologist due to Interminable prostatitis. Nevertheless, just 5 to10% of "prostatitis" cases is really caused by a bacterial contamination.

The purpose was to investigate thoroughly the effect of pumpkin seeds oil phonophoresis among males who are diagnosed with chronic non-bacterial prostatitis.

DETAILED DESCRIPTION:
sixty male outpatients diagnosed with chronic non-bacterial prostatitis. Through sample random sampling procedure the total study population was categorized into three treatment groups; Group A, wherein patients received phonophoresis treatment using pumpkin seeds oil; Group B, where members of the group received trans-perineal continuous low-intensity ultrasound; and Group C, in which the participant received placebo low- intensity ultrasound. All of The three groups of the organized trail received their corresponding treatment daily up-to 3 weeks.

For the analysis participants were recruited from a registry of patients with a diagnosis of CNBP. To be included in the analysis a patient must be evaluated with a confirmed diagnosis. They were examined and diagnosed accordingly by a medical practitioner/urologist.

Patients with concomitant infection, autoimmune diseases, diabetes mellitus, cancer, heart problems/pacemaker, implants (metal, silicone, saline), acute and post-acute injury, thrombophlebitis, impaired sensation, psychiatric diseases, and those with well-known contraindications of ultrasound treatment were excluded from the study. Similarly, those with known hypersensitivity to pumpkin seeds oil and its derivatives, along with those who had received other forms of therapies that could influence the therapeutic outcomes of the study were excluded from the study sample.

ELIGIBILITY:
Inclusion Criteria:

* For the analysis participants were recruited from a registry of patients with a diagnosis of CNBP. To be included in the analysis a patient must be evaluated with a confirmed diagnosis. They were examined and diagnosed accordingly by a medical practitioner/urologist. The patients who were included in the study should have normal laboratory findings

Exclusion Criteria:

* Patients with concomitant infection, autoimmune diseases, diabetes mellitus, cancer, heart problems/pacemaker, implants (metal, silicone, saline), acute and post-acute injury, thrombophlebitis, impaired sensation, psychiatric diseases, and those with well-known contraindications of ultrasound treatment were excluded from the study. Similarly, those with known hypersensitivity to pumpkin seeds oil and its derivatives, along with those who had received other forms of therapies that could influence the therapeutic outcomes of the study were excluded from the study sample.

Ages: 40 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — males with CNBP
Enrollment: 60 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2018-02-19 (Actual)

PRIMARY OUTCOMES:
NIH Chronic Prostatitis Symptom Index (NIH-CPSI) | 3 weeks
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sayed A Tantawy, Study Director — Cairo University
Locations (2):
- Egypt (2):
  - Dr Dalia Kamel, Giza
  - Dr Sayed Tanatwy, Giza

IPD SHARING:
Plan to Share IPD: No